CLINICAL TRIAL: NCT04159298
Title: Novel Multi-planar Neuromuscular Neck Strengthening for the Treatment of Delayed Recovery of Concussion in Adolescence and Young Adults With Cervicogenic Symptoms
Brief Title: Cervicogenic Concussion Rehabilitation With TopSpin360
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Collaborators: TopSpin Technologies Ltd (Industry)
Responsible Party: Principal Investigator, Dr. Lisa Fischer, Director, Sport and Exercise Medicine, Western University, Canada
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CCRT360
Record Dates: First submitted 2019-10-30; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Concussion, Mild
Keywords: rehabilitation; sports medicine; Test a New Treatment; randomized control trial
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group who will undergo the Top Spin 360 study protocol.
  Interventions: Device: Top Spin 360
- Traditional (No Intervention): Control group who undergo traditional usual clinical care comprised of bi-weekly physiotherapy sessions and home-based exercise programs.

INTERVENTIONS:
Device: Top Spin 360 — The TopSpin360 is a dynamic multi-planar neuromuscular training device that has been shown to improve static and dynamic multi-planar neck strength in a healthy athletic population
  Arms: Intervention

SUMMARY:
Concussions occur most frequently in adolescents and often result in significant disruption to daily living for prolonged periods of time. Concussions are an epidemic, with the incidence rates for sports related concussions (SRC) in adolescents up to 0.47 per 1000 athlete exposures. Research would suggest that multi-planar neck strength is a protective factor of SRC risk in adolescents as greater neck strength is associated with a lower SRC risk.(Collins et al) Neck pain is a common symptom associated with SRC that is also associated with prolonged recovery from SRC. (King et al, Van der Naalt et al) Neck pain is also associated with decreased neck muscle strength (DeKoning et al). Our study will address a critical gap in concussion management - multi-planar cervical spine strengthening to specifically rehabilitate the cervicogenic component of prolonged post-concussion symptoms with a cervicogenic component and determine if this approach restores normal neck strength, decreases neck pain and headaches, improves daily global function and allow patients to return to sport and school. work more quickly than those without specific multi-planar neck strengthening.

DETAILED DESCRIPTION:
Overall Design: This will be a randomized clinical trial using a prospective cohort model. A total of 56 adolescents/young adults with concussion symptoms that persist >4 weeks post-trauma and +ve screening for cervical involvement (rated neck pain as a symptom, TOP para cervical or suboccipital spine, +ve cervical flexion-rotation test (Hall et al)) will be assigned randomly into one of two groups: 1) Control group who undergo traditional usual clinical care comprised of bi-weekly physiotherapy sessions and home-based exercise programs (TRADITIONAL), and 2) In combination with standard clinical care as described above, 2 sessions per week training on the TopSpin360 (protocol outlined below). (INTERVENTION). The intervention will last up to 7 weeks or until medical clearance to return to normal daily activities. Balancing as much as possible the impact of age and sport is critical because mechanisms and patterns of injury differ with the patient and the sport in which the concussion occurred. The randomization process will balance the influence of one's sex on the measured outcomes.

Randomization: Patients will be randomized into one of the two groups using a 1:1 ratio to balance recruitment and covariates. A random number generator will be used to assign groups.

Test Sequence: Based on previous work, it is anticipated that 7 weeks of intervention will be required. (Versteegh et al) Following baseline measures (Week 0) upon study entry, tests will be conducted at the midway point (4 weeks) and upon completion (7 weeks) or upon medical clearance to return to sport. The test sessions ideally will occur following the clinical examination with the physician . This will increase convenience for the patient's family who, for this age group, will be with the patient. At each test session a physiotherapist will bring the participant through 1. Cervical Flexion-Rotation test, 2. Deep neck flexor endurance test, 3. a multi-planar static neck strength assessment using a handheld dynamometer (Versteegh et al), 4. Dynamic necks strength assessed via peak RPM and time to complete 20 revolutions clockwise and counterclockwise on the TopSpin360, 5. Joint position error testing (Revel et al), 6. and complete standard questionnaires: SCAT 5 symptom score, Neck Disability Index, Headache Inventory and

Intervention training protocol using TopSpin360: Participants allocated to the INTERVENTION group will participate in 2 training sessions per week using the TopSpin360 neuromuscular neck-training device. Each session will be separated by a minimum of 2 days. Given the target population for this study will include younger subjects than previous training studies using the TopSpin360 and given they will have some neck pathology, a significantly reduced training load (number of revolutions used per set) will be used. The advantage of the TopSpin360 as a training tool is its safety profile in that the device uses self-generated resistance to create the muscular load and training effect.

The attached weight is only 125gm, and the resistance is generated through the centripetal force created as the participant swings the weight about the centrally mounted axis. Much like a hula-hoop, the participant is only capable of spinning the weight as quickly as his or her neck muscles and coordination are capable of getting it spinning, if they fatigue or lose coordination, the weight stops spinning and the resistance is removed. The first 2 weeks will involve 3 sets of 20 revolutions in each direction of clockwise and counterclockwise. Weeks 3 and 4 will involve 3 sets of 30 revolutions in each direction and weeks 4-7 will involve 3 sets of 40 revolutions in each direction.

ELIGIBILITY:
Inclusion Criteria:

* > 28 symptoms cervicogenic symptoms

Exclusion Criteria:

* < 28 symptoms
* no cervicogenic symptoms

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Cervical Flexion-Rotation Test (CFRT) | 8 weeks
  Static neck strength measurement tool
Multi-planar static neck strength (MicroFET2) | 8 weeks
  Dynamic neck strength assessment tool
Deep neck flexor endurance test | 8 weeks
  Timed test to determine how long a participant can hold an isometric contraction of the deep neck flexor

SECONDARY OUTCOMES:
SCAT 5 Symptom Score | 8 weeks
  22 item symptom checklist using a 7 point likert scale from 0 to 6 (0 absence of symptom, 1-2 mild severity, 3-4 moderate severity, 5-6 severe)
Neck Disability Index (NDI) | 8 weeks
  Functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
Headache Disability Inventory (HDI) | 8 weeks
  Consists of 40 items, each requiring a "yes" (four points), "sometimes" (two points), or "no" (zero points) response based on items derived empirically from case history responses of subjects with headache.
Global Disability Index | 8 weeks
  25 item self reported instrument assessing different aspects of disability
SF-36 | 8 weeks
  36-item self-report measure of health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Fowler Kennedy Sports Medicine Clinic, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No